CLINICAL TRIAL: NCT00614965
Title: A Multicenter Randomized Phase II Study of the Combination of Irinotecan/Cisplatin Versus Pemetrexed/Cisplatin as Second-line Treatment of Patients With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: Irinotecan Plus Cisplatin vs Pemetrexed Plus Cisplatin as 2nd Line in NSCLC Stage IIIB/IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: S.Aggelaki, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.16
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Cancer; NSCLC; second-line chemotherapy; irinotecan; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Irinotecan; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IC
  Interventions: Drug: Irinotecan; Drug: Cisplatin
- 2 (Experimental): PC
  Interventions: Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Irinotecan — Irinotecan at the dose of 110 mg/m2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: CPT-11
  Arms: 1
Drug: Cisplatin — Cisplatin at the dose of 80 mg/m2 IV on day 1 every 3 weeks for 6 consecutive cycles
  Other Names: CDDP
Drug: Pemetrexed — Pemetrexed at the dose of 500mg/m2 IV every 3 weeks for 6 consecutive cycles
  Other Names: Alimta
  Arms: 2

SUMMARY:
This trial will compare the efficacy of irinotecan/cisplatin and pemetrexed/cisplatin in the second-line treatment of patients with stage IIIB/IV NSCLC

DETAILED DESCRIPTION:
Non-platinum-based doublets including the newer drugs can be used instead of platinum-based regimens in the first line treatment of patients with advanced NSCLC. Docetaxel or pemetrexed have been proven effective as second-line treatment of patients with NSCLC. In a study conducted by our group the combination of irinotecan/cisplatin demonstrated higher response rates over cisplatin monotherapy in patients progressing after first-line docetaxel/gemcitabine. Moreover, pemetrexed has been combined with the platinums (ie, cisplatin, carboplatin, and oxaliplatin) in NSCLC to yield clinical activity similar to that of other platinum-based doublets. The efficacy of different platinum-based combinations in patients pretreated with non-platinum based first-line chemotherapy is not known.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Age 18 -75 years
* Performance status (WHO) <2
* Patients progressing after first-line docetaxel/gemcitabine treatment
* Adequate bone marrow (absolute neutrophil count >1000/mm3, platelet count >100000/mm3, hemoglobin > 9 gr/ mm3)
* Adequate liver (bilirubin <1.5 times upper limit of normal), renal (Creatinine clearance > 50mg/min) and cardiac (LVEF >50%) function
* Presence of measurable disease (according to RESIST criteria)
* Informed consent

Exclusion Criteria:

* Psychiatric illness or social situation that would preclude study compliance'
* Other concurrent uncontrolled illness.
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Time to Tumor Progression | 1-year
Overall Survival | 1-year
Toxicity profile between the two treatment arms | Toxicity assessment on each chemotherapy cycles
Quality of life assessment | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Aggelaki, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (2):
- Greece (2):
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens

REFERENCES:
- [Derived] Kentepozidis N, Economopoulou P, Christofyllakis C, Chelis L, Polyzos A, Vardakis N, Koinis F, Vamvakas L, Katsaounis P, Kalbakis K, Nikolaou C, Georgoulias V, Kotsakis A. Salvage treatment with irinotecan/cisplatin versus pemetrexed/cisplatin in patients with non-small cell lung cancer pre-treated with a non-platinum-based regimen in the first-line setting: a randomized phase II study of the Hellenic Oncology Research Group (HORG). Clin Transl Oncol. 2017 Mar;19(3):317-325. doi: 10.1007/s12094-016-1532-y. Epub 2016 Aug 4. PMID 27492015